CLINICAL TRIAL: NCT02473393
Title: A Clinical Trial to Assess Three Different Doses of OPS-2071 in Patients With Bacterial Enteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 341-13-002; JapicCTI-152937 (Other: Japic)
Record Dates: First submitted 2015-06-08; First posted 2015-06-16 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Bacterial Enteritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- OPS-2071 50mg/day (Experimental): OPS-2071 50 mg/day：25 mg tablet administered orally twice daily
  Interventions: Drug: OPS-2071 tablet
- OPS-2071 100 mg/day (Experimental): OPS-2071 100 mg/day：50 mg tablet administered orally twice daily
  Interventions: Drug: OPS-2071 tablet
- OPS-2071 200 mg/day (Experimental): OPS-2071 200 mg/day：100 mg tablet administered orally twice daily
  Interventions: Drug: OPS-2071 tablet
- OPS-2071 400 mg/day (Experimental): OPS-2071 400 mg/day：100 mg two tablets administered orally twice daily
  Interventions: Drug: OPS-2071 tablet

INTERVENTIONS:
Drug: OPS-2071 tablet

SUMMARY:
To assess safety, efficacy and pharmacokinetics of multiple dosesin patients with Bacterial Enteritis caused by Clostridium difficile infection(CDI) or Enteric infection.

ELIGIBILITY:
Inclusion Criteria:

* The patient provides written, informed consent before the clinical trial is initiated
* The patient has distinctive symptoms and findings of bacterial enteritis
* The patient has bacterial enteritis with one or more of the following causative pathogens either proven or presumed: C. difficile, Salmonella, Campylobacter, pathogenic E. coli, and other bacteria estimated to cause bacterial enteritis
* The patient and his/her partner are willing to take contraceptive measures from initiation of investigational medicinal products (IMPs) to 4 weeks after administration of IMPs

Exclusion Criteria:

* The patient has severe or progressive underlying disease or complication, making it difficult to ensure safety in the study or proper efficacy assessment
* The patient has a current diagnosis or history of convulsive disorders, such as convulsion and epilepsy
* The patient has a severe hepatic dysfunction
* The patient has a severe cardiac dysfunction
* The patient has cardiac arrhythmia or congenital or sporadic long QTc syndrome. Or the patient is treated with a drug reported to prolong QTc interval
* The patient has a moderate or severe renal dysfunction
* Women with confirmed or suspected pregnancy or breast-feeding women
* Patients judged to be ineligible by the investigator for any other reasons

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-08-20 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshitaka Kotobuki, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (3):
- Kanto, Region, Japan
- Singapore, Singapore
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed as a global trial in Japan, Republic of Korea, and Singapore.
Pre-assignment Details: Subjects with bacterial enteritis were divided into 2 groups, a Clostridium difficile infection (CDI) group for subjects with bacterial enteritis associated with C. difficile infection and an enteric infection (EI) group for subjects with bacterial enteritis for which the causative pathogen was Salmonella, Campylobacter, or pathogenic E. coli. Only one dosage (100 mg) of OPS-2071 was administered to CDI subjects and 3 dosages (100, 50, and 200 mg) were administered to EI subjects.
Groups:
- CDI Group: OPS-2071 was orally administered at a dose of 100 mg twice daily in the morning and evening for 10 days.
- EI Group (50 mg): OPS-2071 was orally administered at a dose of 25 mg twice daily in the morning and evening for 7 days.
  The administration was started with the 100 mg group, and the safety and efficacy during the treatment period were to be assessed by the Data Review Committee. If the 100 mg group had no safety concerns and the efficacy was assessed "effective," 10 subjects each who were not in the 100 mg group were to be randomized to the 200 mg or 50 mg group, and the 2 groups were to be treated in parallel. If the 100 mg group had no safety concerns and the efficacy was assessed "not effective," 10 subjects who were not in the 100 mg group were to be allocated to the 200 mg group as the next step.
- EI Group (100 mg): OPS-2071 was orally administered at a dose of 50 mg twice daily in the morning and evening for 7 days.
  The administration was started with the 100 mg group, and the safety and efficacy during the treatment period were to be assessed by the Data Review Committee. If the 100 mg group had no safety concerns and the efficacy was assessed "effective," 10 subjects each who were not in the 100 mg group were to be randomized to the 200 mg or 50 mg group, and the 2 groups were to be treated in parallel. If the 100 mg group had no safety concerns and the efficacy was assessed "not effective," 10 subjects who were not in the 100 mg group were to be allocated to the 200 mg group as the next step.
- EI Group (200 mg): OPS-2071 was orally administered at a dose of 100 mg twice daily in the morning and evening for 7 days.
  The administration was started with the 100 mg group, and the safety and efficacy during the treatment period were to be assessed by the Data Review Committee. If the 100 mg group had no safety concerns and the efficacy was assessed "effective," 10 subjects each who were not in the 100 mg group were to be randomized to the 200 mg or 50 mg group, and the 2 groups were to be treated in parallel. If the 100 mg group had no safety concerns and the efficacy was assessed "not effective," 10 subjects who were not in the 100 mg group were to be allocated to the 200 mg group as the next step.
Period: Overall Study
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Started | 5 | 12 | 13 | 13
Completed | 5 | 12 | 11 | 12
Not Completed | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all subjects who had received the investigational medicinal product (IMP) at least once and from whom data on at least one efficacy endpoint had been obtained after the start of IMP administration.
Groups:
- Total: Total of all reporting groups
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg) | Total
Number analyzed (Participants) | 5 | 12 | 12 | 12 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 11 | 11 | 12 | 37
  >=65 years | 2 | 1 | 1 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (24.52) | 36.0 (15.78) | 36.3 (16.51) | 35.6 (12.41) | 39.4 (18.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 7 | 5 | 20
  Male | 2 | 7 | 5 | 7 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 4 | 12 | 10 | 10 | 36
  Korean | 0 | 0 | 2 | 1 | 3
  Singaporean | 0 | 0 | 0 | 0 | 0
  Others | 1 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 0 | 0 | 2 | 0 | 2
  Singapore | 1 | 0 | 0 | 0 | 1
  Japan | 4 | 12 | 10 | 12 | 38

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Elimination Rate (BER) in the CDI and EI Groups
Description: Judged according to the assessment criteria for the bacterial strain isolated as the causative pathogen based on the data from the microbiological examination. Analysis was performed by disease group and by dose, and by minimum inhibitory concentration (MIC) values of OPS-2071 for each of the causative strains (Enterotoxigenic E. coli, Enteroaggregative E. coli, Campylobacter sp., C. jejuni, S. aureus, K. oxytoca, and C. perfringens for the EI group). Data were shown as all strains total.
  Concerning microbiological outcome by causative strain, bacteria elimination rate (BER) and its 95% confidence interval (CI) were calculated. The BER was the proportion of causative strains assessed as either "Excellent" or "Good" except for those assessed as "unknown/indeterminate".
Time Frame: CDI group: screening, Day 4 and Day 11 (end of treatment), EI group: screening, Day 4 and Day 8 (end of treatment)
Population: Microbiological per Protocol Set (MPPS) comprised those subjects in the FAS for whom the causative pathogen was identified and for whom microbiological outcome was assessed as "Excellent", "Good", or "Poor" , excluding subjects for whom microbiological outcome was assessed as "unknown/indeterminate".
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 2 | 9 | 9 | 7
percentage of participants | 100.0 [15.8 to 100.0] | 72.7 [39.0 to 94.0] | 90.0 [55.5 to 99.7] | 87.5 [47.3 to 99.7]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of OPS-2071 on Day 4
Description: We measured OPS-2071 concentration in plasma and evaluated Cmax of OPS-2071 in plasma.
Time Frame: Inpatient: 1h, 2h, and 4h after morning administration
Population: Pharmacokinetics Analysis Set (PKS) comprised subjects in whom plasma drug concentration had been measured at least once.
Measure: Mean (Full Range); unit: µg/L
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 1 | 2 | 2 | 2
µg/L | 64 | 29.2 [17.7 to 40.6] | 42.4 [38.5 to 46.2] | 81.9 [62.8 to 101]

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of OPS-2071 on Day 4
Description: We measured OPS-2071 concentration in plasma and evaluated tmax of OPS-2071 in plasma.
Time Frame: 1h, 2h, and 4h after morning administration
Population: as for outcome 2
Measure: Mean (Full Range); unit: h
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 1 | 2 | 2 | 2
h | 4.15 [4.15 to 4.15] | 1.98 [1.95 to 2.00] | 4.08 [4.03 to 4.12] | 2.42 [0.92 to 3.92]

4. Secondary Outcome: The Recurrence Rate of CDI After Multiple Doses of OPS-2071 (for CDI Group Only)
Description: CDI recurrence rate at follow-up (Day 38) or withdrawal was calculated. CDI recurrence rate was the proportion of the subjects judged as "recurrent" against evaluable subjects, except for those with missing data.
Time Frame: Day 38
Population: Clinical per protocol set (CPPS) comprised those subjects in the FAS for whom all scheduled examinations at all specified observation time points up until end of treatment or withdrawal had been performed. Analysis was performed by dose in the proportion of subjects judged as "clinical cure" at end of treatment (EOT) in the CPPS.
Measure: Number; unit: percentage of participants
Arm/Group | CDI Group
Number analyzed (Participants) | 4
percentage of participants | 0.0

5. Secondary Outcome: The Time to Resolution of Diarrhea After Multiple Doses of OPS-2071
Description: The time from the start of dosing until the first formed stool (except in cases where liquid or unformed stools recurred) was evaluated as time to resolution of diarrhea. If formed stool has not been observed, then the subject will be handled as missing data.
Time Frame: CDI group: Day 4, Day 11 (end of treatment) and Day 38, EI group: Day 4 and Day 8 (end of treatment)
Population: CPPS comprised those subjects in the FAS for whom all scheduled examinations at all specified observation time points up until end of treatment or withdrawal had been performed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 3 | 10 | 9 | 9
days | 3.7 (1.53) | 4.3 (1.34) | 4.4 (2.01) | 4.6 (1.42)

6. Secondary Outcome: Stool Frequency Per Day After Multiple Doses of OPS-2071
Description: Under each disease group, the improvement of clinical symptoms (stool frequency/day) were assessed.
Time Frame: CDI group: screening, Day 4, Day 11 (end of treatment) and Day 38, EI group: screening, Day 4 and Day 8 (end of treatment)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: stool frequency/day
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 4 | 10 | 10 | 12
stool frequency/day
  Screening | 5.3 (3.30) | 7.3 (2.91) | 7.1 (2.77) | 9.2 (4.28)
  Day 4 | 1.5 (0.58) | 2.9 (1.52) | 1.4 (0.97) | 2.7 (2.74)
  Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Day 8 |  | 2.0 (1.41) | 1.7 (0.67) | 2.6 (1.93)
  Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Day 11 | 2.3 (0.96) |  |  |
  Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Day 38 | 1.3 (0.58) |  |  |

7. Secondary Outcome: Number of Subjects With Formed Stool, Liquid or Unformed Stool, and Bloody Stool After Multiple Doses of OPS-2071
Description: Under each disease group, the improvement of clinical symptoms ((i.e. formed stool, liquid or unformed stool [3 and more times], and presence of bloody stool) were assessed.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 4 | 10 | 10 | 12
participants
  Formed stool at Screening | 0 | 0 | 0 | 0
  Formed stool on Day 4 | 2 | 7 | 3 | 5
  Formed stool on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Formed stool on Day 8 |  | 7 | 9 | 8
  Formed stool on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Formed stool on Day 11 | 1 |  |  |
  Formed stool on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Formed stool on Day 38 | 2 |  |  |
  Liquid or unformed stool at Screening | 4 | 10 | 10 | 12
  Liquid or unformed stool on Day 4 | 0 | 1 | 0 | 3
  Liquid or unformed stool on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Liquid or unformed stool on Day 8 |  | 0 | 0 | 2
  Liquid or unformed stool on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Liquid or unformed stool on Day 11 | 2 |  |  |
  Liquid or unformed stool on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Liquid or unformed stool on Day 38 | 0 |  |  |
  Bloody stool at Screening | 0 | 2 | 3 | 2
  Bloody stool on Day 4 | 0 | 0 | 0 | 0
  Bloody stool on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Bloody stool on Day 8 |  | 0 | 0 | 0
  Bloody stool on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Bloody stool on Day 11 | 0 |  |  |
  Bloody stool on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Bloody stool on Day 38 | 0 |  |  |

8. Secondary Outcome: Number of Subjects With Abdominal Pain, Nausea, and Vomiting After Multiple Doses of OPS-2071
Description: Under each disease group, he improvement of clinical symptoms (i.e. presence of abdominal pain, nausea, and vomiting) were assessed.
Time Frame: as for outcome 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 4 | 10 | 10 | 12
participants
  Abdominal pain at Screening | 2 | 10 | 10 | 12
  Abdominal pain on Day 4 | 1 | 4 | 3 | 5
  Abdominal pain on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Abdominal pain on Day 8 |  | 1 | 0 | 2
  Abdominal pain on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Abdominal pain on Day 11 | 0 |  |  |
  Abdominal pain on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Abdominal pain on Day 38 | 0 |  |  |
  Nausea at Screening | 1 | 6 | 7 | 2
  Nausea on Day 4 | 0 | 0 | 0 | 0
  Nausea on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Nausea on Day 8 |  | 0 | 0 | 0
  Nausea on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Nausea on Day 11 | 0 |  |  |
  Nausea on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Nausea on Day 38 | 0 |  |  |
  Vomiting at Screening | 0 | 2 | 3 | 0
  Vomiting on Day 4 | 0 | 0 | 0 | 0
  Vomiting on Day 8: number analyzed (Participants) | 0 | 10 | 10 | 12
  Vomiting on Day 8 |  | 0 | 1 | 0
  Vomiting on Day 11: number analyzed (Participants) | 4 | 0 | 0 | 0
  Vomiting on Day 11 | 0 |  |  |
  Vomiting on Day 38: number analyzed (Participants) | 4 | 0 | 0 | 0
  Vomiting on Day 38 | 0 |  |  |

9. Secondary Outcome: Clinical Response Rate (CRR) in the CDI and EI Groups
Description: The CRR and 95% CI at each evaluation time point were calculated. The CRR was calculated as the proportion of the subjects judged as "clinical cure" or "clinical improvement" against evaluable subjects, except for those with missing data.
Time Frame: CDI group: Day 4 and Day 11 (end of treatment), EI group: Day 4 and Day 8 (end of treatment)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
Number analyzed (Participants) | 4 | 10 | 10 | 12
percentage of participants
  Day 4 | 100.0 [39.8 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [73.5 to 100.0]
  End of treatment | 100.0 [39.8 to 100.0] | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7] | 100.0 [73.5 to 100.0]

ADVERSE EVENTS:
Time Frame: From the start day of IMP administration up to Day 38
Description: Adverse events (AEs) occurring after IMP administration were included in assessment of AEs.
  All subjects receiving at least 1 dose of IMP were included in the safety set.
Arm/Group | CDI Group | EI Group (50 mg) | EI Group (100 mg) | EI Group (200 mg)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12 | 1/13 | 0/12
Other Adverse Events (participants affected / at risk) | 3/5 | 4/12 | 8/13 | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CDI Group (N=5) | EI Group (50 mg) (N=12) | EI Group (100 mg) (N=13) | EI Group (200 mg) (N=12)
Pyrexia (General disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CDI Group (N=5) | EI Group (50 mg) (N=12) | EI Group (100 mg) (N=13) | EI Group (200 mg) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-07-15): https://cdn.clinicaltrials.gov/large-docs/93/NCT02473393/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02473393/SAP_001.pdf